CLINICAL TRIAL: NCT00244985
Title: A Phase I/II Pilot Study of the Safety and Efficacy of Rituxan (Chimeric Anti-CD20 Antibody) in Combination With Doxil (Liposomal Doxorubicin) Chemotherapy in Patients With Relapsing or Refractory Indolent or Aggressive B-Cell Lymphoma
Brief Title: Rituximab and Liposomal Doxorubicin in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000447130; RPC 02-04 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent small lymphocytic lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Rituximab and Doxorubicin HCI Liposome (Experimental): Patients receive rituximab IV over 3-8 hours on day 1 and doxorubicin HCl liposome IV over 1-3 hours on day 3
  Interventions: Biological: rituximab; Drug: pegylated liposomal doxorubicin hydrochloride

INTERVENTIONS:
Biological: rituximab — IV
Drug: pegylated liposomal doxorubicin hydrochloride — IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as liposomal doxorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with liposomal doxorubicin may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects of giving rituximab together with liposomal doxorubicin and to see how well they work in treating patients with relapsed or refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety, including qualitative and quantitative toxic effects and their duration and reversibility, of rituximab and doxorubicin HCl liposome in patients with relapsed or refractory, indolent or aggressive CD20-positive B-cell non-Hodgkin's lymphoma.

Secondary

* Determine the efficacy, including overall response rate and durability of objective response, of this regimen in these patients.
* Correlate pretreatment functional, phenotypic, and genotypic characteristics of host immune effector cells with response in patients treated with this regimen.

OUTLINE: This is an open-label, pilot study.

Patients receive rituximab IV over 3-8 hours on day 1 and doxorubicin HCl liposome IV over 1-3 hours on day 3. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 4 years.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following indolent or aggressive B-cell non-Hodgkin's lymphoma (NHL) subtypes:

  * Grade 1-3 follicular lymphoma
  * Mantle cell lymphoma
  * Small lymphocytic lymphoma
  * Diffuse large B-cell lymphoma
  * Diffuse mixed cell lymphoma
  * Marginal zone lymphoma
* Relapsed or refractory CD20-positive disease
* Measurable disease
* Must have received ≥ 1 but < 4 prior standard chemotherapy regimens
* No Burkitt's lymphoma or precursor B-lymphoblastic lymphoma
* No CNS lymphoma

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 6 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin > 7 g/dL

Hepatic

* AST or ALT < 2 times upper limit of normal (unless due to primary disease)
* Bilirubin ≤ 2 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* LVEF ≥ 50% by MUGA and/or 2-D echocardiogram
* No history of New York Heart Association class II-IV cardiac disease
* No congestive heart failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No uncontrolled active bacterial, viral, or fungal infection
* No other serious disease that would preclude study participation
* No other primary malignancy within the past 5 years except squamous cell or basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy
* Prior immunotherapy, including rituximab or other monoclonal antibody, allowed

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy and recovered
* No prior doxorubicin (or equivalent anthracycline) at a cumulative dose > 400 mg/m^2
* No other concurrent chemotherapy

Endocrine therapy

* Nonsteroidal hormones for nonlymphoma-related conditions (e.g., insulin for diabetes) allowed
* No concurrent corticosteroids except for a transient inflammatory reaction (i.e., skin rash or hives)

Radiotherapy

* Recovered from prior radiotherapy
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery (other than diagnostic surgery) and recovered

Other

* No other concurrent antitumor agents
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron S. Czuczman, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Rituximab and Doxorubicin HCI Liposome
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Arm 1: Rituximab and Doxorubicin HCI Liposome
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate at 20 Weeks
Description: Complete Response (CR): During observation no disease is apparent, including measurable and non-measurable disease, for at least 28 days, as confirmed by a second assessment following the original observation of no disease. All nodes visualized on imaging studies or palpable on exams must have regressed to normal size their greatest transverse diameter for nodes > 1.5 em before therapy). Previously involved nodes that were 1.1 to 1.5 in their greatest transverse diameter before treatment must have decreased to 1 cm in their greatest transverse diameter after treatment or by more than 75% in the sum of the products of the greatest diameters (SPD). The patient must also be free from symptoms related to lymphoma, if present before therapy with no worsening in performance status from baseline. Bone marrow, if initially positive at baseline, must be histologically negative for lymphoma and the liver and spleen, if enlarged due to lymphoma at baseline, should be normalized.
Time Frame: 20 weeks
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Rituximab and Doxorubicin HCI Liposome
Number analyzed (Participants) | 42
percentage of participants | 45 [30 to 61]

2. Secondary Outcome: Partial Response Rate at 20 Weeks
Description: Partial Response (PR): A 50% or greater decrease from baseline in the sum of the products of the longest perpendicular diameters of all the measured lesions is noted for at least 28 days as confirmed by a second assessment following the observation of the > or = to 50% decrease. Additionally, no appearance of new lesions is noted.
Time Frame: 20 weeks
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Rituximab and Doxorubicin HCI Liposome
Number analyzed (Participants) | 42
percentage of participants | 19 [9 to 34]

3. Secondary Outcome: Overall Response Rate (Complete and Partial Responses) at 20 Weeks
Description: Complete Response (CR): During observation no disease is apparent, including measurable and non-measurable disease, for at least 28 days, as confirmed by a second assessment following the original observation of no disease. All nodes visualized on imaging studies or palpable on exams must have regressed to normal size their greatest transverse diameter for nodes > 1.5 before therapy. Partial Response (PR): A 50% or greater decrease from baseline in the sum of the products of the longest perpendicular diameters of all the measured lesions is noted for at least 28 days as confirmed by a second assessment following the observation of the > or = to 50% decrease. Additionally, no appearance of new lesions is noted.
Time Frame: 20 weeks
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Rituximab and Doxorubicin HCI Liposome
Number analyzed (Participants) | 42
percentage of participants | 64 [48 to 78]

4. Secondary Outcome: Progression Free Survival (PFS) Rate at 2 Years
Description: Progressive disease is defined as at least a 20% increase in the sum of the longest diameter of target lesions or the appearance of new lesions.
Time Frame: 2 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Rituximab and Doxorubicin HCI Liposome
Number analyzed (Participants) | 42
percentage of participants | 42 [32 to 62]

5. Secondary Outcome: Overall Survival (OS) Rate at 2 Years
Description: Overall survival was defined as time from date of treatment initiation until date of death due to any cause.
Time Frame: 2 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Rituximab and Doxorubicin HCI Liposome
Number analyzed (Participants) | 42
percentage of participants | 83 [68 to 92]

ADVERSE EVENTS:
Arm/Group | Arm 1: Rituximab and Doxorubicin HCI Liposome
Serious Adverse Events (participants affected / at risk) | 6/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Rituximab and Doxorubicin HCI Liposome (N=42)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (3)
Mucosal infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Rituximab and Doxorubicin HCI Liposome (N=42)
Anemia (Blood and lymphatic system disorders) | 10 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (18)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (4)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (9)
Tinnitus (Ear and labyrinth disorders) | 1 (17)
Conjunctivitis (Eye disorders) | 1 (32)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (31)
Anal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (31)
Dysphagia (Gastrointestinal disorders) | 2 (8)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (18)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 7 (11)
Vomiting (Gastrointestinal disorders) | 1 (20)
Chills (General disorders) | 9 (10)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 18 (25)
Fever (General disorders) | 5 (6)
Flu like symptoms (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (3)
Infusion related reaction (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (3)
Localized edema (General disorders) | 2 (3)
Pain (General disorders) | 8 (35)
Bronchial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 5 (6)
Mucosal infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (2)
Papulopustular rash (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (8)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (11)
tooth infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (6)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (10)
Investigations - Other, specify (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 16 (16)
Platelet count decreased (Investigations) | 19 (20)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (57)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (32)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (15)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (18)
Dizziness (Nervous system disorders) | 1 (17)
Dysgeusia (Nervous system disorders) | 1 (21)
Headache (Nervous system disorders) | 1 (37)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (5)
Depression (Psychiatric disorders) | 1 (31)
Insomnia (Psychiatric disorders) | 1 (17)
Restlessness (Psychiatric disorders) | 1 (14)
Bladder spasm (Renal and urinary disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (11)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (23)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 30 (47)
Hypertension (Vascular disorders) | 1 (35)
Hypotension (Vascular disorders) | 1 (24)
Superior vena cava syndrome (Vascular disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes